CLINICAL TRIAL: NCT03166306
Title: Angiogenic Imaging in Pulmonary Arterial Hypertension
Acronym: AIPAH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Paul B Yu, Physician; Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017P000249
Record Dates: First submitted 2017-05-09; First posted 2017-05-25 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Arterial Hypertension; Exercise Associated Pulmonary Arterial Hypertension
Keywords: pulmonary vascular disease; pulmonary vascular imaging
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: The investigators propose to enroll 10 patients with known severe idiopathic or familial PAH, 10 individuals with exercise-associated PAH (EPAH), felt to be a milder and early stage of PAH, and 10 healthy volunteers with no evidence of cardiopulmonary disease. Baseline PET-CT scans will be obtained 7 days after the injection of [89Zr]-bevacizumab. Follow- up imaging will be obtained 12 months status post enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Patients with idiopathic or familial PAH (Experimental): Ten patients with severe idiopathic or familial PAH will undergo PET-CT imaging with [89Zr]-bevacizumab.
  Interventions: Diagnostic Test: PET-CT Imaging with [89Zr]-bevacizumab
- Patients with exercise associated PAH (Experimental): Ten patients with exercise associated PAH (EPAH) will undergo PET-CT imaging with [89Zr]-bevacizumab.
  Interventions: Diagnostic Test: PET-CT Imaging with [89Zr]-bevacizumab
- Healthy volunteers (Active Comparator): Ten individuals with no known cardiopulmonary disease will undergo PET-CT imaging with [89Zr]-bevacizumab.
  Interventions: Diagnostic Test: PET-CT Imaging with [89Zr]-bevacizumab

INTERVENTIONS:
Diagnostic Test: PET-CT Imaging with [89Zr]-bevacizumab — Subjects will receive 1 millicurie of 89Zr and less than 5 mg of bevacizumab, followed by PET-CT imaging.

SUMMARY:
Pulmonary arterial hypertension (PAH) is a disorder of elevated pulmonary vascular resistance characterized by progressive remodeling and obliteration of vessels of the distal pulmonary circulation. Outcomes in PAH could be improved with earlier diagnosis, and with the early deployment of therapies before irreversible changes have occurred. This study tests the sensitivity of positron emission tomography (PET)-CT scanning with [89Zr]-bevacizumab, a radioisotope-conjugated anti-VEGF antibody for detecting pulmonary vascular remodeling in PAH disease. This test could enable non-invasive diagnosis early in the course of the disease, and potentially improve outcomes in PAH,

DETAILED DESCRIPTION:
PAH is a disease of progressive remodeling and obliteration of the distal pulmonary vasculature. The overexpression of VEGF-A in the pulmonary vasculature of patients with PAH and animal models of disease is thought to reflect a process of disordered angiogenesis that is tightly coupled to disease progression. It is hypothesized that positron emission tomography (PET)-CT scan utilizing [89Zr]-bevacizumab, a radioisotope-conjugated humanized monoclonal antibody against VEGF-A, would provide a sensitive and specific molecular imaging modality to detect pulmonary vascular remodeling activity.

To test this hypothesis the investigators propose a Phase I/II pilot study to enroll 10 patients with known severe idiopathic or familial PAH, 10 individuals with exercise-associated PAH (EPAH), thought to be a mild and early stage of PAH, and 10 healthy volunteers with no evidence of cardiopulmonary disease. This pilot study will compare standardized uptake values (SUV) for the retention of [89Zr]-bevacizumab in the distal pulmonary vasculature in these three populations. The kinetics of equilibration and wash-out of this probe will be assessed with sequential scans at 4 and 7 days following the injection of radionuclide. In patients with PAH or EPAH, repeat scans will be performed 1 year after the initial scan to assess whether changes in clinical status correlate with [89Zr]-bevacizumab retention.

The ability of these protocols to discriminate between the lungs of healthy individuals versus patients with PAH or EPAH will be evaluated using the measure of peripheral lung tissue probe SUV, corresponding to distal pulmonary vessel uptake, normalized to the proximal aortic SUV, corresponding to the blood pool. These data will be used to define normative values for healthy controls versus PAH patients, and to generate cutoffs in signaling ratios with optimal sensitivity and specificity for disease detection. These normative ranges will be applied to the EPAH cohort to determine if this test retains sensitivity and specificity for a potentially milder, earlier form of PAH.

This study is divided into 4 Aims:

AIM 1: Test the hypothesis that expression of VEGF-A discerned by [89Zr]-bevacizumab imaging is increased in the distal pulmonary vascular bed in PAH patients compared to healthy individuals.

AIM 2: Test the hypothesis that expression of VEGF-A discerned by [89Zr]-bevacizumab imaging is increased in the distal pulmonary vascular bed in patients with exercise-associated PAH compared to healthy individuals.

AIM 3: Ascertain whether or not distal pulmonary vascular uptake of [89Zr]-bevacizumab correlates with clinical markers of PAH severity, including 6 minute walk distance, New York Heart Association functional class, right atrial pressure, mean pulmonary artery pressure, pulmonary vascular resistance, cardiac index, NT-proBNP, tricuspid annular plane systolic excursion (TAPSE) by echocardiography.

AIM 4: Ascertain whether or not changes in distal pulmonary vascular uptake of [89Zr]-bevacizumab over 1 year in patients with PAH or EPAH correlates with changes in clinical status based on clinical markers of PAH severity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at screening;
* Documented diagnosis Group 1 PAH confirmed by resting mean pulmonary artery pressure greater than 25 mm of Hg, pulmonary vascular resistance greater than 3 Wood units, and pulmonary wedge pressure less than 12 mm of Hg measured by right heart catheterization at the time of diagnosis and before initiation of PAH specific therapy clinically stable for 60 or more days prior to enrollment, defined as no changes in medical regimen and no hospitalizations;
* Prior diagnosis of exercise-associated PAH (EPAH) confirmed by normal resting hemodynamics (mean pulmonary artery pressure < 25 mm of Hg, pulmonary artery wedge pressure < 12 mm of Hg, and pulmonary vascular resistance < 3 Wood units) measured by right heart catheterization at rest and abnormal hemodynamic response to exercise characterized by increase in mean pulmonary artery pressure > 30 mm Hg, pulmonary artery wedge pressure < 20 mm Hg, and pulmonary vascular resistance > 1 Wood unit at peak exercise and cardiac output less than 10 L/min before initiation of any PAH specific therapy. Patients need to be clinically stable for 60 or more days prior to enrollment, defined as no changes in medical regimen and no hospitalizations;
* Willingness to participate as evidenced by signing of the informed consent;

Exclusion Criteria:

* Prior history of chronic infectious disease, tuberculosis, or severe fungal disease; chronic hepatitis B or C infection; renal insufficiency; interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis; known chronic pericardial effusion, pleural effusion, or ascites; chronic liver disease; myeloproliferative disorders in the past 5 years; non-basal cell malignancy or treated lymphoproliferative disease within the past 5 years; known HIV positive; life expectancy of <3 years;
* Chronic inflammatory condition such as lupus or rheumatoid arthritis, ulcerative colitis or Crohn's disease;
* White blood cell count <2,500/uL, hematocrit < 30 percent, or platelet count < 50,000/uL;
* Elevated liver transaminase levels (AST or ALT) 20 % above upper limit of normal (ULN) or albumin 20 % below the lower limit of normal (LLN);
* Creatinine clearance < 45 mL/min as estimated with the Cockroft-Gault equation;
* Women who are pregnant or breastfeeding;
* Men or women who plan to have children during the study period or who are unwilling to use effective forms of contraception;
* Known active cancer;
* Chronic use of oral steroid therapy or other immunosuppressive or biologic response modifiers (see Exclusionary Medication List in Manual of Operations). Eligible study participants will be encouraged to have up to date pneumococcal and influenza vaccinations as recommended based on their age and underlying medical conditions;
* Evidence of interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis in the past 12 months by chest X-ray. For participants who have not had a chest X-ray during the 12 months prior to enrollment in the study, a chest X-ray will be obtained at baseline as part of the study protocol;
* New York Heart Association Class IV congestive heart failure;
* Severe asthma or COPD defined by FEV1 less than 50% predicted and FEV1/FVC less than 70% per PFTs in the past 12 months;
* Active tobacco use during the prior 10 years;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Distal pulmonary SUV of [89Zr]-bevacizumab | Baseline measurement at entry into study
  PET-CT measurement of standardized uptake values (SUV) for retention of [89Zr]-bevacizumab in peripheral lung tissues, normalized to proximal aortic retention corresponding to the blood pool.

SECONDARY OUTCOMES:
Change in distal pulmonary SUV of [89Zr]-bevacizumab | Measurement at 12 months following initial measurement
  Change in PET-CT measurement of standardized uptake values (SUV) for retention of [89Zr]-bevacizumab in peripheral lung tissues, normalized to proximal aortic retention corresponding to the blood pool, compared over a 12 month interval.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Yu, MD PhD, Principal Investigator — Brigham and Women's Hospital; Aaron B Waxman, MD PhD, Principal Investigator — Brigham and Women's Hospital; Marcelo F Di Carli, MD, Principal Investigator — Brigham and Women's Hospital; Ivana Nikolic, MD, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make individual participant data available to other researchers, outside of the publication of datasets in peer-reviewed literature.